CLINICAL TRIAL: NCT06056089
Title: Safety Efficacy, and Cost-effectiveness of Modified Doses of Ready-to-use Therapeutic and Supplementary Foods for the Treatment of Moderate Acute Malnutrition Among Children 6-59 Months of Age in Ethiopia
Brief Title: Modified Dosage for Moderate Acute Malnutrition (MODAM-MAM)
Acronym: MODAM-MAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Action Against Hunger USA (Other)
Collaborators: University of Washington (Other); Ethiopian Public Health Institute (Other Government)
Responsible Party: Principal Investigator, Heather Stobaugh, Senior Research and Learning Specialist, Action Against Hunger USA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MODAM-MAM
Record Dates: First submitted 2023-09-08; First posted 2023-09-28 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Moderate Acute Malnutrition

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): 1 sachet (535 kcal) of RUSF per day
  Interventions: Dietary Supplement: ready-to-use supplementary food (RUSF)
- MAM Experimental A (Experimental): 1 sachet (500 kcal) of RUTF per day
  Interventions: Dietary Supplement: ready-to-use therapeutic food (RUTF)
- MAM Experimental B (Experimental): 2 sachets (1000 kcal) of RUTF per day
  Interventions: Dietary Supplement: ready-to-use therapeutic food (RUTF)

INTERVENTIONS:
Dietary Supplement: ready-to-use supplementary food (RUSF) — standard formulation meeting UNICEF specifications: https://www.unicef.org/supply/media/16636/file/S0000248-RUSF-Specification.pdf
  Arms: Control Group
Dietary Supplement: ready-to-use therapeutic food (RUTF) — standard formulation meeting UNICEF specifications: https://www.unicef.org/supply/sites/unicef.org.supply/files/2023-04/U239977-RUTF-Novel-Specification.pdf
  Arms: MAM Experimental A; MAM Experimental B

SUMMARY:
Protocols for the community-based management of acute malnutrition (CMAM) have not changed significantly for more than 20 years, with relatively complex treatment protocols and persistent supply chain challenges that have limited overall program coverage, leaving millions of malnourished children without care annually. The overarching goal of this research project is to simultaneously test two novel simplified approaches in CMAM with potential to improve program coverage. The simplified approach includes two parallel clinical trials for SAM and MAM treatment. Two fixed-dose regimes of RUTF will be tested against the current fixed-dose regimen of RUSF for children with MAM.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-59 months
2. Reside in the catchment area of the health post where the trial is to be conducted without plans to leave the area over the next year
3. Uncomplicated moderate acute malnutrition, as defined by no signs of severe illness that would require referral to inpatient facility
4. Pass appetite test conducted at the time of enrollment
5. Consent for randomization into the study given by mother, father, and/or other primary caregiver
6. Mid-upper arm circumference of 115-124 mm without nutritional edema
7. Weight-for-height Z-score (WHZ) between -2 and -3

Exclusion Criteria:

1. Complicated acute malnutrition with severe illness requiring transfer to a stabilization center or hospital for treatment. This includes, but is not limited to: a. Hypothermia b. High fever c. Signs of hypoglycemia d. Lethargy or altered mental status e. Moderate to severe dehydration f. Shock g. Other medical complications requiring hospitalization or higher-level medical evaluation
2. Treatment for acute malnutrition, either as an inpatient or outpatient, within the past 3 months
3. Known chronic medical illness such as severe cerebral palsy, severe congenital anomalies such as unrepaired congenital heart disease, Down syndrome, hydrocephalus, unrepaired cleft lip or palate, or other conditions that would be expected to contribute to difficulty feeding the prescribed amounts of therapeutic or supplementary food

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2400 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
short-term nutritional recovery from MAM | up to 16 weeks
  two consecutive weeks with MUAC > 12.4 cm and/or WHZ >= -2, depending on enrollment criteria

SECONDARY OUTCOMES:
weight gain during treatment | weekly for up to 16 weeks
mid-upper-arm circumference (MUAC) gain during treatment | weekly for up to 16 weeks
length/height gain during treatment | weekly for up to 16 weeks
changes to phase angle (PhA) as measured by bioelectrical impedance analysis | up to weekly for up to 16 weeks
changes to extracellular water (ECW) as measured by bioelectrical impedance analysis | up to weekly for up to 16 weeks
changes to total body water (TBW) as measured by bioelectrical impedance analysis | up to weekly for up to 16 weeks
changes to fat free mass as measured by bioelectrical impedance analysis | up to weekly for up to 16 weeks
changes in immunological function during treatment as measured by quantification of T-cell recombination excision circles (TRECs) and kappa-deleting recombination excision circles (KRECs) on dried blood spots | up to weekly for up to 16 weeks
rates of acute illness, including diarrhea, vomiting, and fever during treatment | weekly for up to 16 weeks
mortality rate | weekly for up to 16 weeks
hospitalization rate | weekly for up to 16 weeks
duration of treatment required prior to short-term recovery | weekly for up to 16 weeks
medium-term mortality rate | up to 6 months post-recovery
  calculated as number of children who die divided by total number of children initially enrolled
medium-term rate of development of acute malnutrition | up to 6 months post-recovery
  calculated as number of children who develop acute malnutrition by the total number of children initially enrolled
medium-term rates of relapse to SAM | up to 6 months post-recovery
medium-term rates of relapse to MAM | up to 6 months post-recovery
medium-term rates of hospitalization | up to 6 months post-recovery
medium-term weight gain | 6 months post-recovery
medium-term MUAC gain | 6 months post-recovery
medium-term length/height gain | 6 months post-recovery
medium-term phase angle (PhA) as measured by bioelectrical impedance analysis | 6 months post-recovery
medium-term extracellular water (ECW) as measured by bioelectrical impedance analysis | 6 months post-recovery
medium-term total body water (TBW) as measured by bioelectrical impedance analysis | 6 months post-recovery
medium-term fat free mass as measured by bioelectrical impedance analysis | 6 months post-recovery
medium-term immunological function during treatment as measured by quantification of T-cell recombination excision circles (TRECs) and kappa-deleting recombination excision circles (KRECs) on dried blood spots | 6 months post-recovery
short-term cost-efficiency | up to 16 weeks
  calculated as the total costs of the treatment for all children divided by the number of children who achieve nutritional recovery
medium-term cost-efficiency | 6 months post-recovery
  calculated as the total costs of the treatment for all children divided by the number of children who sustain nutritional recovery

CONTACTS AND LOCATIONS:
Overall Officials: Heather C Stobaugh, Principal Investigator — Action Against Hunger USA; Indi Trehan, Principal Investigator — University of Washington; Yosef B Asefaw, MSc, Principal Investigator — Ethiopian Public Health Institute
Locations (3):
- Ethiopia (3):
  - Sekota, Sekota, Amhara
  - Teltele, Teltelē, Oromiya
  - Gode, Gode, Somali

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Trehan I, Beyene Y, Darsene H, Adams BS, Wrabel M, Gizaw G, Legese LA, Cichon B, Chitekwe S, Shellemew MW, Tessema M, Stobaugh HC. The Modified Dosages for Acute Malnutrition (MODAM) study: protocol for three integrated randomized controlled trials of novel approaches for the management of childhood wasting in Ethiopia. BMC Nutr. 2025 Apr 8;11(1):71. doi: 10.1186/s40795-025-01054-w. PMID 40200326